CLINICAL TRIAL: NCT00633594
Title: Phase I/II Study Evaluating Rituximab, Lenalidomide, and Bortezomib in the First-Line or Second-Line Treatment of Patients With Mantle Cell Lymphoma
Brief Title: Rituximab, Lenalidomide, and Bortezomib in Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 58
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; Rituximab; Lenalidomide; Bortezomib; Phase 1/2
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Bortezomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab/bortezomib/lenalidomide (Experimental): Patients in Phase I & II to receive treatment with rituximab, bortezomib and lenalidomide in 21-day cycles up to 6 cycles.
  Phase I: Cohorts of 3 patients will be enrolled at escalating dose levels to determine the maximum tolerated dose (MTD). Doses may be de-escalated if necessary.
  Phase II: patients will be treated with the MTD determined in Phase I.
  Interventions: Drug: Rituximab; Drug: Bortezomib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Rituximab — DL 1, DL 2, and DL 3: 375 mg/m2 IV Days 1, 8, and 15; Cycles 2-6: 375 mg/m2 IV Day 1
  Same for DL-1.
  Other Names: Rituxan; MabThera
Drug: Bortezomib — DL 1, DL 2, and DL 3: 1.3 mg/m2 IV Days 1, 4, 8, and 11
  Same for DL-1.
  Other Names: Velcade
Drug: Lenalidomide — DL 1: 15 mg PO daily Days 1-14 followed by 7 days of rest
  DL 2: 20 mg PO daily Days 1-14 followed by 7 days of rest
  DL 3: 25 mg PO daily Days 1-14 followed by 7 days of rest
  DL-1: 10 mg PO daily Days 1-14 followed by 7 days of rest
  Other Names: Revlimid

SUMMARY:
This is a Phase I/II multicenter, open-label, dose-escalation study of rituximab, bortezomib, and lenalidomide in the first-line or second-line treatment of patients with Mantle Cell Lymphoma (MCL).

DETAILED DESCRIPTION:
The combination of lenalidomide with bortezomib has not been studied in patients with MCL, but feasibility and tolerability has been demonstrated in patients with multiple myeloma. Thus, almost every 2-drug combination of rituximab, lenalidomide, and bortezomib has been tested, or is being tested. We hypothesize that all three drugs are important in MCL, and therefore propose to combine all 3 agents (rituximab, bortezomib, and lenalidomide) in a schedule that is convenient to lymphoma patients.

Approximately 18 patients may be enrolled in the Phase I portion of the study. Approximately 45 patients are planned for enrollment in Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. All study participants must be registered into the Mandatory Revlimid Risk Evaluation and Mitigation Strategies (REMS) Program, and be willing and able to comply with the requirements of the REMS program.
2. Histology: biopsy-proven mantle cell lymphoma (MCL).
3. Prior therapy: both newly diagnosed patients and relapsed or refractory patients who have received one prior therapy are eligible. Patients who have previously received high-dose chemotherapy with peripheral stem cell support are eligible.
4. Presence of at least one lymph node evaluable or mass measurable for response.
5. Platelets ≥ 75,000/µL and absolute neutrophil count (ANC) ≥ 1,000/µL within 14 days of study registration (unless the treating physician deems the neutropenia is related to bone marrow involvement, then an ANC of > 750/mm3 is allowed).
6. Renal function assessed by calculated creatinine clearance between ≥ 30 ml/min and ˂60ml/min by the Cockcroft-Gault method within 14 days of study registration
7. Total bilirubin ≤ 1.5x upper limit of normal (ULN), aspartate transaminase (AST) (SGOT) and alanine transaminase (ALT) (SGOT) ≤ 3 x ULN
8. Eastern Cooperative Oncology Group (ECOG) performance of 0, 1, or 2.
9. Recovery from any previous treatment therapy.
10. Females of childbearing potential (FCBP) must adhere to the scheduled pregnancy testing required in the Revlimid REMS® program, must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior and again within 24 hours of starting lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by Revlimid REMS Program) and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
11. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of Revlimid REMS® program.
12. Ability to understand and willingness to voluntarily sign a written informed consent document before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

1. Patient has >1.5 x ULN total bilirubin.
2. Peripheral neuropathy ≥ CTCAE grade 2.
3. Relapsed or refractory patients who have received more than one prior therapy.
4. Pregnant or breastfeeding females. (Lactating females must agree not to breastfeed while taking lenalidomide.)
5. Female patients who have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on Day 1 before first dose of study drug, if applicable.
6. Thrombolic or embolic events (such as a cerebrovascular accident, including transient ischemic attacks) within the past 6 months.
7. Pulmonary hemorrhage/bleeding event ≥ CTCAE grade 2 within 28 days of the first dose of study drug.
8. Any other hemorrhage/bleeding event ≥ CTCAE grade 3 ≤ 28 days of the first dose of study drug
9. Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
10. Central nervous system (CNS) involvement by lymphoma at time of enrollment.
11. Other medical conditions or psychiatric illness that would potentially interfere with patient participation in this trial.
12. A second malignancy, other than basal cell carcinoma of the skin or in situ carcinoma of the cervix, unless the tumor was treated with curative intent at least 2 years previously.
13. Previous evidence of hypersensitivity to bortezomib, boron, mannitol, thalidomide, (and development of erythema nodosum if characterized by a desquamating rash), or rituximab (true anaphylaxis, not a rituximab-infusion reaction).
14. Known human immunodeficiency virus (HIV) infection or chronic hepatitis A, B, or C. Patients who are HIV positive or who are positive for chronic hepatitis A, B, or C will be excluded due to increased risk for bone marrow suppression and other toxicities.
15. Active, clinically serious infection > CTCAE grade 2. Patients may be eligible upon resolution of the infection.
16. Evidence or history of bleeding diathesis or coagulopathy.
17. Major surgery, open biopsy, or significant traumatic injury within 28 days of the first dose of study drug.
18. Use of any other standard chemotherapy, radiation therapy, or experimental drug for the treatment of MCL within 28 days of starting treatment.
19. Any condition that impairs a patient's ability to swallow whole pills. Impairment of gastrointestinal function (GI) or GI disease that may significantly alter the absorption of lenalidomide (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
20. Patients with grade 3/4 cardiac problems, as defined by the New York Heart Association (NYHA) criteria or any of the following:

    * History of uncontrolled or symptomatic angina
    * History of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation
    * Myocardial infarction < 6 months from study entry
    * Uncontrolled or symptomatic congestive heart failure
    * Ejection fraction below the institutional normal limit
    * Electrocardiographic evidence of acute ischemia or active conduction system
    * Any other cardiac condition that, in the opinion of the treatment physician, would make this protocol unreasonably hazardous for the patient
    * Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
21. Uncontrolled hypertension (systolic blood pressure [BP] > 180 or diastolic BP > 100mm Hg) or uncontrolled cardiac arrhythmias.
22. Any prior use of lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-06; Primary Completion 2015-04 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian W Flinn, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Providence Medical Group, Terre Haute, Indiana
  - RHHP/ Hope Cancer Center, Terre Haute, Indiana
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosch F, Lopez-Guillermo A, Campo E, Ribera JM, Conde E, Piris MA, Vallespi T, Woessner S, Montserrat E. Mantle cell lymphoma: presenting features, response to therapy, and prognostic factors. Cancer. 1998 Feb 1;82(3):567-75. doi: 10.1002/(sici)1097-0142(19980201)82:33.0.co;2-z. PMID 9452276
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Corral LG, Haslett PA, Muller GW, Chen R, Wong LM, Ocampo CJ, Patterson RT, Stirling DI, Kaplan G. Differential cytokine modulation and T cell activation by two distinct classes of thalidomide analogues that are potent inhibitors of TNF-alpha. J Immunol. 1999 Jul 1;163(1):380-6. PMID 10384139
- [Background] Davies FE, Raje N, Hideshima T, Lentzsch S, Young G, Tai YT, Lin B, Podar K, Gupta D, Chauhan D, Treon SP, Richardson PG, Schlossman RL, Morgan GJ, Muller GW, Stirling DI, Anderson KC. Thalidomide and immunomodulatory derivatives augment natural killer cell cytotoxicity in multiple myeloma. Blood. 2001 Jul 1;98(1):210-6. doi: 10.1182/blood.v98.1.210. PMID 11418482
- [Background] Dredge K, Horsfall R, Robinson SP, Zhang LH, Lu L, Tang Y, Shirley MA, Muller G, Schafer P, Stirling D, Dalgleish AG, Bartlett JB. Orally administered lenalidomide (CC-5013) is anti-angiogenic in vivo and inhibits endothelial cell migration and Akt phosphorylation in vitro. Microvasc Res. 2005 Jan;69(1-2):56-63. doi: 10.1016/j.mvr.2005.01.002. PMID 15797261
- [Background] Ghielmini M, Schmitz SF, Cogliatti S, Bertoni F, Waltzer U, Fey MF, Betticher DC, Schefer H, Pichert G, Stahel R, Ketterer N, Bargetzi M, Cerny T; Swiss Group for Clinical Cancer Research. Effect of single-agent rituximab given at the standard schedule or as prolonged treatment in patients with mantle cell lymphoma: a study of the Swiss Group for Clinical Cancer Research (SAKK). J Clin Oncol. 2005 Feb 1;23(4):705-11. doi: 10.1200/JCO.2005.04.164. Epub 2004 Dec 14. PMID 15598978
- [Background] Howard OM, Gribben JG, Neuberg DS, Grossbard M, Poor C, Janicek MJ, Shipp MA. Rituximab and CHOP induction therapy for newly diagnosed mantle-cell lymphoma: molecular complete responses are not predictive of progression-free survival. J Clin Oncol. 2002 Mar 1;20(5):1288-94. doi: 10.1200/JCO.2002.20.5.1288. PMID 11870171
- [Background] Kaufman DS, Lewis RL, Hanson ET, Auerbach R, Plendl J, Thomson JA. Functional endothelial cells derived from rhesus monkey embryonic stem cells. Blood. 2004 Feb 15;103(4):1325-32. doi: 10.1182/blood-2003-03-0799. Epub 2003 Oct 16. PMID 14563647
- [Background] Lenz G, Dreyling M, Hoster E, Wormann B, Duhrsen U, Metzner B, Eimermacher H, Neubauer A, Wandt H, Steinhauer H, Martin S, Heidemann E, Aldaoud A, Parwaresch R, Hasford J, Unterhalt M, Hiddemann W. Immunochemotherapy with rituximab and cyclophosphamide, doxorubicin, vincristine, and prednisone significantly improves response and time to treatment failure, but not long-term outcome in patients with previously untreated mantle cell lymphoma: results of a prospective randomized trial of the German Low Grade Lymphoma Study Group (GLSG). J Clin Oncol. 2005 Mar 20;23(9):1984-92. doi: 10.1200/JCO.2005.08.133. Epub 2005 Jan 24. PMID 15668467
- [Background] Moreau P, Pylypenko H, Grosicki S, Karamanesht I, Leleu X, Grishunina M, Rekhtman G, Masliak Z, Robak T, Shubina A, Arnulf B, Kropff M, Cavet J, Esseltine DL, Feng H, Girgis S, van de Velde H, Deraedt W, Harousseau JL. Subcutaneous versus intravenous administration of bortezomib in patients with relapsed multiple myeloma: a randomised, phase 3, non-inferiority study. Lancet Oncol. 2011 May;12(5):431-40. doi: 10.1016/S1470-2045(11)70081-X. Epub 2011 Apr 18. PMID 21507715
- [Background] Romaguera JE, Fayad L, Rodriguez MA, Broglio KR, Hagemeister FB, Pro B, McLaughlin P, Younes A, Samaniego F, Goy A, Sarris AH, Dang NH, Wang M, Beasley V, Medeiros LJ, Katz RL, Gagneja H, Samuels BI, Smith TL, Cabanillas FF. High rate of durable remissions after treatment of newly diagnosed aggressive mantle-cell lymphoma with rituximab plus hyper-CVAD alternating with rituximab plus high-dose methotrexate and cytarabine. J Clin Oncol. 2005 Oct 1;23(28):7013-23. doi: 10.1200/JCO.2005.01.1825. Epub 2005 Sep 6. PMID 16145068
- [Background] Weisenburger DD, Sanger WG, Armitage JO, Purtilo DT. Intermediate lymphocytic lymphoma: immunophenotypic and cytogenetic findings. Blood. 1987 Jun;69(6):1617-21. PMID 3555648
- [Background] Foran JM, Rohatiner AZ, Cunningham D, Popescu RA, Solal-Celigny P, Ghielmini M, Coiffier B, Johnson PW, Gisselbrecht C, Reyes F, Radford JA, Bessell EM, Souleau B, Benzohra A, Lister TA. European phase II study of rituximab (chimeric anti-CD20 monoclonal antibody) for patients with newly diagnosed mantle-cell lymphoma and previously treated mantle-cell lymphoma, immunocytoma, and small B-cell lymphocytic lymphoma. J Clin Oncol. 2000 Jan;18(2):317-24. doi: 10.1200/JCO.2000.18.2.317. PMID 10637245
- [Background] Schafer PH, Gandhi AK, Loveland MA, Chen RS, Man HW, Schnetkamp PP, Wolbring G, Govinda S, Corral LG, Payvandi F, Muller GW, Stirling DI. Enhancement of cytokine production and AP-1 transcriptional activity in T cells by thalidomide-related immunomodulatory drugs. J Pharmacol Exp Ther. 2003 Jun;305(3):1222-32. doi: 10.1124/jpet.102.048496. Epub 2003 Mar 20. PMID 12649301

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Lenalidomide 15mg PO QD: Cycle 1: rituximab 375 mg/m2 intravenously (IV) on Days 1, 8, and 15; bortezomib 1.3 mg/ m2 subcutaneously (SC) on Days 1, 4, 8, and 11; and lenalidomide 15 mg by mouth (PO) daily on Days 1-14. Cycles 2 - 6: rituximab 375 mg/m2 IV on Day 1; bortezomib 1.3 mg/ m2 SC on Days 1, 4, 8, and 11; and lenalidomide 15 mg PO daily on Days 1-14.
- Phase I - Lenalidomide 10mg PO QD; Phase II - Lenalidomide 10mg PO QD: Cycle 1: rituximab 375 mg/m2 intravenously (IV) on Days 1, 8, and 15; bortezomib 1.3 mg/ m2 subcutaneously (SC) on Days 1, 4, 8, and 11; and lenalidomide 10 mg by mouth (PO) daily on Days 1-14. Cycles 2 - 6: rituximab 375 mg/m2 IV on Day 1; bortezomib 1.3 mg/ m2 SC on Days 1, 4, 8, and 11; and lenalidomide 10 mg PO daily on Days 1-14.
Period: Overall Study
Arm/Group | Phase I - Lenalidomide 15mg PO QD | Phase I - Lenalidomide 10mg PO QD | Phase II - Lenalidomide 10mg PO QD
Started | 5 | 8 | 26
Completed | 5 | 3 | 16
Not Completed | 0 | 5 | 10
Not completed — Adverse Event | 0 | 4 | 7
Not completed — Death | 0 | 1 | 2
Not completed — Disease Progression | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Based on efficacy evaluable population, all participants that received any study therapy. Participants were stratified based on phase of study (Phase I vs Phase II) and previous treatment status prior to study start (Previously Untreated vs Previously Treated (relapsed or refractory))
Groups:
- Phase I - Lenalidomide 15mg PO QD: Cycle 1: rituximab 375 mg/m2 intravenously (IV) on Days 1, 8, and 15; bortezomib 1.3 mg/ m2 subcutaneously (SC) on Days 1, 4, 8, and 11; and lenalidomide 15 mg by mouth (PO) daily on Days 1-14. Cycles 2 - 6: rituximab 375 mg/m2 IV on Day 1; bortezomib 1.3 mg/ m2 SC on Days 1, 4, 8, and 11; and lenalidomide 15 mg PO daily on Days 1 14. .
- Phase I - Lenalidomide 10mg PO QD; Phase II - Lenalidomide 10mg PO QD: Cycle 1: rituximab 375 mg/m2 intravenously (IV) on Days 1, 8, and 15; bortezomib 1.3 mg/ m2 subcutaneously (SC) on Days 1, 4, 8, and 11; and lenalidomide 10 mg by mouth (PO) daily on Days 1-14. Cycles 2 - 6: rituximab 375 mg/m2 IV on Day 1; bortezomib 1.3 mg/ m2 SC on Days 1, 4, 8, and 11; and lenalidomide 10 mg PO daily on Days 1 14.
- Total: Total of all reporting groups
Arm/Group | Phase I - Lenalidomide 15mg PO QD | Phase I - Lenalidomide 10mg PO QD | Phase II - Lenalidomide 10mg PO QD | Total
Number analyzed (Participants) | 5 | 8 | 26 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 7 | 12
  >=65 years | 2 | 6 | 19 | 27
Age, Continuous [Median (Full Range); unit: years] | 60 [52 to 70] | 69 [60 to 80] | 69 [55 to 88] | 69 [52 to 88]
Age, Customized [Count of Participants; unit: Participants]
  Previously Treated : <= 18 years | 0 | 0 | 0 | 0
  Previously Treated : Between 18 and 65 years | 3 | 0 | 0 | 3
  Previously Treated : >= 65 years | 1 | 1 | 5 | 7
  Previously Untreated : <= 18 years | 0 | 0 | 0 | 0
  Previously Untreated : Between 18 and 65 years | 0 | 2 | 7 | 9
  Previously Untreated : >= 65 years | 1 | 5 | 14 | 20
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender based on participants' previous treatment prior to initiating study treatment (previously treated and previously untreated)
  Participants
    Previously Treated : Female | 1 | 1 | 2 | 4
    Previously Treated : Male | 3 | 0 | 3 | 6
    Previously Untreated : Female | 0 | 1 | 5 | 6
    Previously Untreated : Male | 1 | 6 | 16 | 23
Gender [Count of Participants; unit: Participants]
  Female | 1 | 2 | 7 | 10
  Male | 4 | 6 | 19 | 29
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 26 | 39
Previous Treatment for Mantle Cell Lymphoma (MCL) [Number; unit: participants] — Includes participants with relapsed or refractory MCL who have received one previous treatment prior to starting study treatment, and those with previously untreated MCL prior to starting study treatment.
  participants
    Previously Untreated | 1 | 7 | 21 | 29
    Previously Treated | 4 | 1 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Lenalidomide Combined With Bortezomib and Rituximab in Phase I Participants
Description: Determination of the maximum tolerated dose (MTD) of lenalidomide combined with bortezomib and rituximab, defined as the highest dose at which ≤1 of 6 patients experiences a dose-limiting toxicity according to the NCI CTCAE v. 4.03.
  MTD of Lenalidomide was tested, included with 1.3 mg/m2 subcutaneous (D1, 4, 8, 11) bortezomib, 375 mg/m2 (D1, 8, 15 of Cycle 1, D1 on subsequent cycles) rituximab.
  Three dose limiting toxicities were reported in two patients (grade 4 neutropenia and grade 3 neuropathy, grade 3 rash)
Time Frame: Collected from day of first dose to the end of the first treatment cycle, up to 21 days
Population: Includes patients that were enrolled in both lenalidomide dose levels (10 mg PO daily, 15 mg PO daily) in the Phase I portion of the study
Measure: Number; unit: mg lenalidomide, orally, daily, day 1-14
Groups:
- Phase I Participants (10 mg/15 mg Lenalidomide): Cycle 1: rituximab 375 mg/m2 intravenously (IV) on Days 1, 8, and 15; bortezomib 1.3 mg/ m2 subcutaneously (SC) on Days 1, 4, 8, and 11; and lenalidomide 10 or 15 mg by mouth (PO) daily on Days 1-14. Cycles 2 - 6: rituximab 375 mg/m2 IV on Day 1; bortezomib 1.3 mg/ m2 SC on Days 1, 4, 8, and 11; and lenalidomide 10 or 15 mg PO daily on Days 1-14.
  Includes participants tested on two separate dose levels, 15 mg by mouth (PO) daily (5 participants) or 10 mg PO daily (8 participants)
Arm/Group | Phase I Participants (10 mg/15 mg Lenalidomide)
Number analyzed (Participants) | 13
mg lenalidomide, orally, daily, day 1-14 | 10

2. Primary Outcome: Incidence of Non-Serious Adverse Events as a Measure of Safety and Tolerability, Phase II
Description: A count of affected participants with non-serious adverse events (regardless of relationship to study treatments) occurring in >= 15% of treated patients enrolled in the Phase II section of the study.
  Lenalidomide DL-1 dose (10 mg orally, once daily (PO QD)) Day 1-14 followed by 7 days of rest, Rituximab 375 mg/m2 IV Days 1, 8, and 15 of Cycle 1; Cycles 2-6: 375 mg/m2 IV Day 1, Bortezomib 1.3 mg/m2 subcutaneous Days 1, 4, 8, and 11 for Cycles 1-6
Time Frame: Collected from day of first dose to 30 days after the last dose of study medication, a maximum of 18 weeks and 30 days after last study treatment
Population: Includes patients that were enrolled in the Phase II section of the study
Measure: Number; unit: participants
Groups:
- Phase II - Lenalidomide 10mg PO QD: Lenalidomide DL-1 dose (10 mg orally, once daily (PO QD)) Day 1-14 followed by 7 days of rest, Rituximab 375 mg/m2 IV Days 1, 8, and 15 of Cycle 1; Cycles 2-6: 375 mg/m2 IV Day 1, Bortezomib 1.3 mg/m2 IV Days 1, 4, 8, and 11 for Cycles 1-6
Arm/Group | Phase II - Lenalidomide 10mg PO QD
Number analyzed (Participants) | 26
participants
  Rash | 19
  Fatigue | 18
  Thrombocytopenia | 16
  Leukopenia | 13
  Nausea | 12
  Diarrhea | 11
  Edema | 11
  Hyperglycemia | 11
  Peripheral Neuropathy | 10
  Neutropenia | 10
  Hypoalbuminemia | 10
  Constipation | 9
  Hypocalcemia | 9
  Pain in Extremity | 9
  Anemia | 8
  Cough | 8
  Fever | 8
  Dehydration | 7
  Pruritus | 7
  Dyspnea | 7
  Hyponatremia | 7
  Insomnia | 6
  Abdominal Pain | 6
  Dizziness | 6
  Hypokalemia | 6
  Weight Loss | 6
  Anorexia | 5
  Erythema | 5
  Hypomagnesemia | 5
  Allergic Reaction | 5
  Chills | 5
  Hyperhidrosis | 5
  Myalgia | 4
  Headache | 4
  Mucositis | 4
  Hypoglycemia | 4

3. Secondary Outcome: Overall Response Rate (ORR) of Phase I and Phase II Participants
Description: Response to treatment (Complete Response (CR) or Partial Response (PR)) determined using Non-Hodgkin's Lymphoma Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007.) CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms; PR: 50% or greater decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or extranodal masses, no increase in the size of other nodes, liver or spleen, no new sites of disease, patients who achieve CR but have persistent morphologic bone marrow involvement; Stable Disease (SD): failing to attain PR or CR, but not fulfilling criteria for progressive disease; Progressive Disease (PD)/Relapse: appearance of new lesions more than 1.5 cm in any axis, 50% or greater increase from nadir SPD of any previously involved sites, 50% or greater increase in the longest diameter of any single previously identified node or extranodal mass more than 1 cm in short axis.
Time Frame: Every 6 weeks until treatment discontinuation then every 3 months thereafter, projected average 24 months
Population: The efficacy evaluable population (all participants who have received any study treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Participants (10 mg Lenalidomide): Cycle 1: rituximab 375 mg/m2 intravenously (IV) on Days 1, 8, and 15; bortezomib 1.3 mg/ m2 subcutaneously (SC) on Days 1, 4, 8, and 11; and lenalidomide 10 mg by mouth (PO) daily on Days 1-14. Cycles 2 - 6: rituximab 375 mg/m2 IV on Day 1; bortezomib 1.3 mg/ m2 SC on Days 1, 4, 8, and 11; and lenalidomide 10 mg PO daily on Days 1-14.
Arm/Group | Phase I Participants (10 mg/15 mg Lenalidomide) | Phase II Participants (10 mg Lenalidomide)
Number analyzed (Participants) | 13 | 26
Participants | 12 | 21

4. Secondary Outcome: Overall Response Rate (ORR) of Previously Treated and Previously Untreated Participants
Description: as for outcome 3
Time Frame: Every 6 weeks until treatment discontinuation then every 3 months thereafter, projected average 24 months
Population: The efficacy evaluable population (all participants who have received any study treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Previously Treated Participants: The efficacy evaluable population (all patients who have received any study treatment) in Phase I and Phase II of the study who were refractory to/relapsed from their previous treatment.
  Includes 4 participants in Phase I - Lenalidomide15 mg PO QD, 1 participant in Phase I - Lenlidomide10 mg PO QD and 5 participants in Phase II - Lenalidomide 10 mg PO QD
- Previously Untreated Participants: The efficacy evaluable population (all patients who have received any study treatment) in Phase I and Phase II of the study who not received any previous treatment prior to initiating study treatment.
  Includes 1 participant in Phase I - Lenalidomide15 mg PO QD, 7 participants in Phase I - Lenlidomide10 mg PO QD and 21 participants in Phase II - Lenalidomide 10 mg PO QD
Arm/Group | Previously Treated Participants | Previously Untreated Participants
Number analyzed (Participants) | 10 | 29
Participants | 8 | 25

5. Secondary Outcome: Time to Best Response of Phase I and Phase II Participants
Description: Measured from the time of study entry to the documented beginning of response (CR or PR). This is measured in responders per Non-Hodgkin's Lymphoma Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007.) CR: complete disappearance of detectable clinical evidence of disease and disease-related symptoms; PR: 50% or greater decrease in sum of product of diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase in size of other nodes, liver or spleen, no new disease sites, patients with CR and persistent morphologic bone marrow involvement.
  Time to Best Response will be examined using time-to-event analysis methods. Kaplan-Meier figures will be generated and the log-rank test will be used to examine differences existing between various levels of stratification.
Time Frame: Every 3 months (+/- 2 weeks) after discontinuation of study treatment for 2 years
Population: All participants that received study treatment that were evaluable for a response assessment (one participant in Phase I and two participants in Phase II were considered unevaluable, discontinuing prior to first post-baseline response assessment)
Measure: Median (Full Range); unit: days
Arm/Group | Phase I Participants (10 mg/15 mg Lenalidomide) | Phase II Participants (10 mg Lenalidomide)
Number analyzed (Participants) | 12 | 24
days | 63.50 [59.00 to 169.00] | 71.50 [47.00 to 523.00]

6. Secondary Outcome: Time to Best Response of Previously Treated and Previously Untreated Participants
Description: Measured from the time of study entry to the documented beginning of response (CR or PR). This is measured in responders per Non-Hodgkin's Lymphoma Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007.) CR: complete disappearance of detectable clinical evidence of disease and disease-related symptoms; PR: 50% or greater decrease in sum of product of diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase in size of other nodes, liver or spleen, no new disease sites, patients with CR and persistent morphologic bone marrow involvement.
Time Frame: Every 3 months (+/- 2 weeks) after discontinuation of study treatment for 2 years
Population: All patients that received study treatment that were evaluable for a response assessment (2 previously untreated participants and 1 previously treated participant were considered unevaluable, discontinuing prior to first post-baseline response assessment)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Previously Treated Participants | Previously Untreated Participants
Number analyzed (Participants) | 10 | 29
months | 2.04 [1.5441 to 4.2710] | 2.37 [2.0370 to 4.2053]

7. Secondary Outcome: Duration of Response (DoR) of Phase I and Phase II Participants
Description: Measured from the documented beginning of response (CR or PR) to the time of relapse. This is measured in responders per Non-Hodgkin's Lymphoma Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007.) CR: complete disappearance of detectable clinical evidence of disease and disease-related symptoms; PR: 50% or greater decrease in sum of product of diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase in size of other nodes, liver or spleen, no new disease sites, patients with CR and persistent morphologic bone marrow involvement.
  Duration of Response will be examined using time-to-event analysis methods. Kaplan-Meier figures will be generated and the log-rank test will be used to examine differences existing between various levels of stratification.
Time Frame: Every 3 months (+/- 2 weeks) after discontinuation of study treatment for 2 years or until documented disease progression
Population: All participants that received study treatment that were responders (achieved a PR or better)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase I Participants (10 mg/15 mg Lenalidomide): Cycle 1: rituximab 375 mg/m2 intravenously (IV) on Days 1, 8, and 15; bortezomib 1.3 mg/ m2 subcutaneously (SC) on Days 1, 4, 8, and 11; and lenalidomide 10 or 15 mg by mouth (PO) daily on Days 1-14. Cycles 2 - 6: rituximab 375 mg/m2 IV on Day 1; bortezomib 1.3 mg/ m2 SC on Days 1, 4, 8, and 11; and lenalidomide 10 or 15mg PO daily on Days 1-14.
  Includes participants tested on two separate dose levels, 15 mg by mouth (PO) daily (5 participants) or 10 mg PO daily (8 participants)
Arm/Group | Phase I Participants (10 mg/15 mg Lenalidomide) | Phase II Participants (10 mg Lenalidomide)
Number analyzed (Participants) | 12 | 21
months | 25.72 [5.3224 to 52.665] | 17.81 [4.6982 to 21.092]

8. Secondary Outcome: Duration of Response (DoR) of Previously Treated and Previously Untreated Participants
Description: Measured from the documented beginning of response (CR or PR) to the time of relapse. This is measured in responders per Non-Hodgkin's Lymphoma Revised Response Criteria for Malignant Lymphoma (Cheson et al. 2007.) CR: complete disappearance of detectable clinical evidence of disease and disease-related symptoms; PR: 50% or greater decrease in sum of product of diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase in size of other nodes, liver or spleen, no new disease sites, patients with CR and persistent morphologic bone marrow involvement.
Time Frame: as for outcome 7
Population: All participants that received study treatment that were responders (achieved a PR or better)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Previously Treated Participants | Previously Untreated Participants
Number analyzed (Participants) | 8 | 25
months | 17.94 [2.8583 to 46.982] | 21.09 [5.6509 to 52.665]

9. Secondary Outcome: Progression Free Survival (PFS) of Phase I and Phase II Participants
Description: Defined as the time from entry onto study until lymphoma progression or death from any cause.
  Progression Free Survival will be examined using time-to-event analysis methods. Kaplan-Meier figures will be generated and the log-rank test will be used to examine differences existing between various levels of stratification.
Time Frame: Every 3 months (+/- 2 weeks) after discontinuation of study treatment for 2 years, then every 6 months after documented disease progression
Population: All participants that received study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Participants (10 mg/15 mg Lenalidomide) | Phase II Participants (10 mg Lenalidomide)
Number analyzed (Participants) | 13 | 26
months | 27.70 [7.2608 to 55.097] | 19.35 [7.5236 to 25.298]

10. Secondary Outcome: Progression Free Survival (PFS) of Previously Treated and Previously Untreated Participants
Description: as for outcome 9
Time Frame: as for outcome 9
Population: All participants that received study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Previously Treated Participants | Previously Untreated Participants
Number analyzed (Participants) | 10 | 29
months | 12.4517 [0.4271 to 27.6632] | 25.2649 [7.4908 to 60.4189]

11. Secondary Outcome: Overall Survival of Phase I and Phase II Participants
Description: Defined as the date of study entry to the date of death.
  Overall Survival will be examined using time-to-event analysis methods. Kaplan-Meier figures will be generated and the log-rank test will be used to examine differences existing between various levels of stratification
Time Frame: as for outcome 9
Population: all participants that received study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Participants (10 mg/15 mg Lenalidomide) | Phase II Participants (10 mg Lenalidomide)
Number analyzed (Participants) | 13 | 26
months | 51.45 [21.520 to 71.294] | 35.35 [22.374 to NA] — Not applicable (N/A) was reported as the maximum of the 95% confidence interval due to having insufficient data to provide the upper confidence limit estimate

12. Secondary Outcome: Overall Survival of Previously Treated and Previously Untreated Participants
Description: as for outcome 11
Time Frame: as for outcome 9
Population: all participants that received study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Previously Treated Participants | Previously Untreated Participants
Number analyzed (Participants) | 10 | 29
months | 28.4189 [0.4271 to 51.4168] | 71.2608 [35.3183 to 71.2608]

ADVERSE EVENTS:
Time Frame: 8 years
Description: Time frame from the initiation of study treatment for the first patient enrolled until all patients off-treatment into the survival follow-up interval
Groups:
- Phase I - Lenalidomide 15mg PO QD: Cycle 1: rituximab 375 mg/m2 intravenously (IV) on Days 1, 8, and 15; bortezomib 1.3 mg/ m2 subcutaneously (SC) on Days 1, 4, 8, and 11; and lenalidomide 15 mg by mouth (PO) daily on Days 1-14. Cycles 2 - 6: rituximab 375 mg/m2 IV on Day 1; bortezomib 1.3 mg/ m2 SC on Days 1, 4, 8, and 11; and lenalidomide 15 mg PO daily on Days 1 14.
Arm/Group | Phase I - Lenalidomide 15mg PO QD | Phase I - Lenalidomide 10mg PO QD | Phase II - Lenalidomide 10mg PO QD
Serious Adverse Events (participants affected / at risk) | 2/5 | 6/8 | 13/26
Other Adverse Events (participants affected / at risk) | 5/5 | 8/8 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Lenalidomide 15mg PO QD (N=5) | Phase I - Lenalidomide 10mg PO QD (N=8) | Phase II - Lenalidomide 10mg PO QD (N=26)
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 1
Acute Renal Failure (Renal and urinary disorders) | 0 | 0 | 1
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 1 | 0
Clostridium Difficile (Infections and infestations) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 2
Gastrointestinal- Intussusception (Gastrointestinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Infection- Lung (Pneumonia) (Infections and infestations) | 0 | 1 | 2
Infection- Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Infection- Septic Shock (Infections and infestations) | 0 | 1 | 0
Infection- Varicella (Infections and infestations) | 0 | 0 | 2
Infection- Viral Syndrome (Infections and infestations) | 0 | 1 | 0
Mental Status Change (Psychiatric disorders) | 0 | 0 | 1
Opioid Withdrawal (General disorders) | 0 | 0 | 1
Pain- Non Cardiac Chest (General disorders) | 0 | 0 | 1
Pain- NOS (General disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Platelet Count Decreased (Blood and lymphatic system disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Secondary Malignancy- Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Lenalidomide 15mg PO QD (N=5) | Phase I - Lenalidomide 10mg PO QD (N=8) | Phase II - Lenalidomide 10mg PO QD (N=26)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 6
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 3
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 2
ALLERGIC REACTION (Immune system disorders) | 0 | 0 | 5
ALLERGIC REACTION (INSECT BITE) (Immune system disorders) | 0 | 1 | 0
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
ANEMIA (Blood and lymphatic system disorders) | 1 | 2 | 8
ANOREXIA (Metabolism and nutrition disorders) | 1 | 2 | 5
ANXIETY (Psychiatric disorders) | 2 | 2 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 3
ASTHENIA (General disorders) | 0 | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
BENIGN PROSTATE HYPERPLASIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BLURRED VISION (Eye disorders) | 0 | 0 | 2
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0
CHEST CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
CHEST PAIN (General disorders) | 0 | 0 | 2
CHILLS (General disorders) | 0 | 0 | 5
CONSTIPATION (Gastrointestinal disorders) | 1 | 3 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 8
CREATININE LEVELS DECREASED (Investigations) | 0 | 0 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 3 | 7
DEPRESSION (Psychiatric disorders) | 1 | 2 | 2
DESQUAMATION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DIABETES (Metabolism and nutrition disorders) | 0 | 1 | 0
DIARRHEA (Gastrointestinal disorders) | 2 | 4 | 11
DIZZINESS (Nervous system disorders) | 1 | 1 | 6
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 3
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 2 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 2
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7
EDEMA (General disorders) | 1 | 3 | 11
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 5
ESOPHAGITIS (Gastrointestinal disorders) | 0 | 1 | 0
EYELID DYSFUNCTION (Eye disorders) | 0 | 1 | 0
FATIGUE (General disorders) | 5 | 7 | 18
FEVER (General disorders) | 0 | 2 | 8
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 2
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 1
HEADACHE (Nervous system disorders) | 1 | 1 | 4
HEART FAILURE (Cardiac disorders) | 0 | 1 | 0
HEMATOCRIT DECREASED (Investigations) | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 1 | 3
HOT FLASHES (General disorders) | 0 | 0 | 3
HYPERBILIRUBINEMIA (Hepatobiliary disorders) | 0 | 0 | 3
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1 | 11
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 | 0 | 3
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 | 0 | 3
HYPERTENSION (Vascular disorders) | 1 | 1 | 3
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 0 | 1 | 10
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 | 1 | 9
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 | 0 | 4
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 | 1 | 6
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 | 0 | 5
HYPONATREMIA (Metabolism and nutrition disorders) | 0 | 0 | 7
HYPOTENSION (Vascular disorders) | 1 | 3 | 3
HYPOTHERMIA (General disorders) | 0 | 1 | 0
INFECTION (Infections and infestations) | 0 | 0 | 3
INSOMNIA (Nervous system disorders) | 1 | 3 | 6
INVOLUNTARY MOVEMENTS (Nervous system disorders) | 0 | 2 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 13
MOOD ALTERATION (Psychiatric disorders) | 0 | 0 | 2
MUCOSITIS (Gastrointestinal disorders) | 0 | 1 | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
NASAL DRAINAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
NAUSEA (Gastrointestinal disorders) | 1 | 5 | 12
NEURALGIA (Nervous system disorders) | 0 | 0 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 4 | 10
ORAL PAIN (Gastrointestinal disorders) | 0 | 1 | 1
PAIN (General disorders) | 0 | 1 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
PERIPHERAL NEUROPATHY (Nervous system disorders) | 5 | 5 | 10
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 4 | 7
RASH (Skin and subcutaneous tissue disorders) | 3 | 5 | 19
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 2
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
SINUS INFECTION (Infections and infestations) | 0 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 2
SORE THROAT (Gastrointestinal disorders) | 0 | 0 | 2
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 1 | 0
STOMACH PAIN (Gastrointestinal disorders) | 1 | 0 | 2
SYNCOPE (Nervous system disorders) | 0 | 1 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 2
TASTE ALTERATION (Nervous system disorders) | 2 | 3 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 4 | 16
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 | 1 | 1
TREMOR (Nervous system disorders) | 0 | 0 | 3
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 | 1 | 3
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0
URINARY TRACT INFECTION (Renal and urinary disorders) | 0 | 1 | 1
URINARY TRACT PAIN (Renal and urinary disorders) | 0 | 1 | 0
URINE DISCOLORATION (Renal and urinary disorders) | 0 | 1 | 0
VAGINAL INFECTION (Infections and infestations) | 0 | 1 | 0
VISION CHANGE (Eye disorders) | 0 | 0 | 2
VOMITING (Gastrointestinal disorders) | 0 | 2 | 3
WATERING EYES (Eye disorders) | 1 | 0 | 0
WEIGHT LOSS (Investigations) | 1 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.